CLINICAL TRIAL: NCT00107198
Title: Treatment of Children With Newly-Diagnosed Low Stage Lymphocyte Predominant Hodgkin Disease (LPHD)
Brief Title: Treating Young Patients With Newly Diagnosed, Low Stage, Lymphocyte Predominant Hodgkin Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHOD03P1; NCI-2009-00376 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AHOD03P1; CDR0000419921; COG-AHOD03P1; AHOD03P1 (Other: Children's Oncology Group); AHOD03P1 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Ann Arbor Stage I Childhood Hodgkin Lymphoma; Ann Arbor Stage II Childhood Hodgkin Lymphoma; Childhood Nodular Lymphocyte Predominant B-Cell Lymphoma
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Vincristine

ARMS (1):
- Treatment (surgery, combination chemotherapy, radiotherapy) (Experimental): COMBINATION CHEMOTHERAPY: Patients receive doxorubicin hydrochloride IV over 10-30 minutes and cyclophosphamide IV over 1 hour on day 1, vincristine IV over 1 minute on days 1 and 8, and prednisone PO or IV two or three times daily on days 1-7. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve CR after 3 courses of therapy proceed to follow-up. Patients who do not achieve a CR proceed to involved-field radiotherapy.
  IFRT: Beginning within 3 weeks after completion of combination chemotherapy, patients undergo IFRT once daily, 5 days a week for 2.8 weeks (14 treatments).
  Interventions: Procedure: Conventional Surgery; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Prednisone; Radiation: Radiation Therapy; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Conventional Surgery — Undergo surgery
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Prednisone — Given IV or PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Radiation: Radiation Therapy — Undergo IFRT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This clinical trial is studying how well surgery and/or combination chemotherapy with or without radiation therapy or observation only work in treating young patients with newly diagnosed stage I or stage II lymphocyte predominant Hodgkin disease (LPHD). Surgery may be an effective treatment for LPHD. Drugs used in chemotherapy, such as doxorubicin, vincristine, prednisone, and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill cancer cells. Giving more than one drug (combination chemotherapy) with or without radiation therapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To preserve the excellent cure rate in patients with lymphocyte predominant Hodgkin disease (LPHD) while employing a treatment strategy that minimizes the exposure to chemotherapy and radiation therapy in appropriate patients.

II. To estimate the proportion of stage I patients (with a single involved lymph node that is totally resected) who can be cured with surgery alone.

III. To estimate the proportions of stage I unresected, stage I resected (whose disease has recurred after observation), and stage II LPHD patients who can be cured with adriamycin (doxorubicin)/vincristine/prednisone/cyclophosphamide (AV-PC) x 3, with involved field radiation therapy (IFRT) for those who are not in a CR after chemotherapy.

IV. To reduce the potential for long-term toxicity of LPHD treatment.

OUTLINE: This is a pilot study.

Patients with stage IA disease who underwent confirmed complete resection of a single involved lymph node at diagnosis undergo observation only*.

Patients with stage IA disease who underwent possible complete resection of a single involved lymph node at diagnosis undergo imaging at 6-7 weeks after surgery. Patients with a confirmed complete resection by imaging undergo observation only*. Patients who do not demonstrate complete resection by imaging proceed to combination chemotherapy with or without radiotherapy.

Patients with stage IA disease who underwent a fine needle aspiration of a single involved lymph node OR an incomplete resection of a single involved lymph node at diagnosis may undergo a second surgery to achieve complete resection. Patients who undergo complete resection during the second surgery undergo imaging at 6-7 weeks after surgery. Patients with a confirmed complete resection by imaging undergo observation only*. Patients who do not undergo a second surgery OR do not achieve complete resection with the second surgery proceed to combination chemotherapy with or without radiotherapy. Patients with stage IA disease with involvement of more than 1 lymph node OR stage IIA disease proceed directly to combination chemotherapy with or without radiotherapy.

NOTE: *Patients with recurrent disease after observation only undergo biopsy and restaging and then proceed to combination chemotherapy with or without radiotherapy. (AS OF AMENDMENT #4, THE TREATMENT ARM FOR PATIENTS WHOSE CANCER RECURRED AFTER OBSERVATION ALONE IS NOW CLOSED)

COMBINATION CHEMOTHERAPY: Patients receive doxorubicin hydrochloride intravenously (IV) over 10-30 minutes and cyclophosphamide IV over 1 hour on day 1, vincristine IV over 1 minute on days 1 and 8, and prednisone orally (PO) or IV two or three times daily on days 1-7. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) after 3 courses of therapy proceed to follow-up. Patients who do not achieve a CR proceed to involved-field radiotherapy.

INVOLVED-FIELD RADIOTHERAPY (IFRT): Beginning within 3 weeks after completion of combination chemotherapy, patients undergo IFRT once daily, 5 days a week for 2.8 weeks (14 treatments).

Patients are followed every 3 months for 2 years, every 6 months for 3 years, annually for 5 years, and then every 5 years for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, previously untreated, biopsy-proven lymphocyte predominant Hodgkin disease (LPHD) are eligible for this protocol as follows:

  * Diagnosis of LPHD must be made using the Revised European American Lymphoma (REAL)/World Health Organization (WHO) classification criteria and will be confirmed by rapid pathology central review
  * Clinical stages as follows:

    * Stage IA without bulk disease
    * Stage IIA without bulk disease
  * Patients with "B" symptoms or bulk disease are NOT eligible for this study
* Slides for rapid central pathology review must be sent to the Biopathology Center (BPC)
* Serum glutamic oxalo-acetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 times upper limit of normal (ULN)
* Total bilirubin =< 1.5 times ULN
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min
* Creatinine based on age/gender as follows:

  * No greater than 0.4 mg/dL (for patients 1 to 5 months of age)
  * No greater than 0.5 mg/dL (for patients 6 to 11 months of age)
  * No greater than 0.6 mg/dL (for patients 1 year of age)
  * No greater than 0.8 mg/dL (for patients 2 to 5 years of age)
  * No greater than 1.0 mg/dL (for patients 6 to 9 years of age)
  * No greater than 1.2 mg/dL (for patients 10 to 12 years of age)
  * No greater than 1.4 mg/dL (for female patients >= 13 years of age)
  * No greater than 1.5 mg/dL (for male patients 13 to 15 years of age)
  * No greater than 1.7 mg/dL (for male patients >= 16 years of age)
* Shortening fraction of >= 27% by echocardiogram or ejection fraction of >= 50% by multigated radionuclide angiogram (MUGA)
* Lactating females must agree that they will not breastfeed a child if they are to receive chemotherapy or radiation treatment*
* Female patients of childbearing potential must have a negative pregnancy test if they are to receive chemotherapy or radiation treatment*
* Males and females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method if they are to receive chemotherapy or radiation treatment*
* Note: *Pregnant or breastfeeding women with stage I, single involved lymph node and confirmed (by Quality Assurance Review Center [QARC ]) total resection, are eligible for the observation arm only; no chemotherapy or radiation treatment will be administered to pregnant or breastfeeding women
* No prior chemotherapy
* More than 30 days since prior systemic corticosteroids
* No prior radiotherapy
* All patients and/or their parents or legal guardians must sign a written informed consent

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2006-01-02 (Actual); Primary Completion 2015-10-06 (Actual); Study Completion 2030-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Burton E Appel, Principal Investigator — Children's Oncology Group
Locations (170):
- United States (147):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Cabell-Huntington Hospital, Huntington, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Schneider Children's Medical Center of Israel, Petah Tikua, Israel
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgery or Combination Chemotherapy, With/Without Radiotherapy: Patients receive doxorubicin hydrochloride 50 mg/m2 IV over 10-30 minutes and cyclophosphamide 800 mg/mg2 IV over 1 hour on day 1, vincristine sulfate 1.4 mg/m2 IV (2.8 mg maximum) over 1 minute on days 1 and 8, and prednisone 40 mg/m2/day PO or IV two or three times daily on days 1-7. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve CR after 3 courses of therapy proceed to follow-up. Patients who do not achieve a CR proceed to involved-field radiation therapy (IFRT).
  IFRT: Beginning within 3 weeks after completion of combination chemotherapy, patients undergo IFRT once daily, 5 days a week for 2.8 weeks (14 treatments).
  doxorubicin hydrochloride: Given IV
  conventional surgery: Undergo surgery
  cyclophosphamide: Given IV
  prednisone: Given IV or PO
  vincristine sulfate: Given IV
  radiation therapy: Undergo IFRT
Period: Overall Study
Arm/Group | Surgery or Combination Chemotherapy, With/Without Radiotherapy
Started | 188
Completed | 136
Not Completed | 52
Not completed — Lack of Efficacy | 28
Not completed — Lost to Follow-up | 12
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 6
Not completed — Ineligible | 5

BASELINE CHARACTERISTICS:
Arm/Group | Surgery or Combination Chemotherapy, With/Without Radiotherapy
Number analyzed (Participants) | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 184
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 13 [4 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 164
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 21
  White | 144
  More than one race | 0
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  Canada | 20
  United States | 162
  Israel | 2
  Australia | 2
  Puerto Rico | 2

OUTCOME MEASURES:

1. Primary Outcome: Failure-free Survival (FFS)
Description: The time to a treatment (strategy) failure, where failure includes one of the following occurrences as a first event: disseminated disease (> Stage I/II) progression or recurrence at any time, local disease progression or recurrence anytime during or after treatment with AV-PC +/- IFRT, occurrence of a second malignant neoplasm, death from any cause.
Time Frame: At 5 years
Population: Of 188 patients enrolled, five ineligible patients and five patients who did not receive the upfront chemotherapy +/- RT per protocol were excluded from this analysis. 178 patients are included. The median follow-up for the 164 censored patients is 61.2 (range 3.5-107.4) months.
Measure: Number (95% Confidence Interval); unit: Probability participants
Arm/Group | Surgery or Combination Chemotherapy, With/Without Radiotherapy
Number analyzed (Participants) | 178
Probability participants | 0.91 [0.86 to 0.95]

2. Secondary Outcome: Event-free Survival
Description: Failure includes one of the following occurrences as a first event: relapse/progression or second malignancy from enrollment.
Time Frame: At 5 years
Population: Of 188 patients enrolled, five ineligible patients were excluded from this analysis. 183 patients are included. The median follow-up time for the 155 censored patients is 61.2 months (range 0.03-107.4).
Measure: Number (95% Confidence Interval); unit: Probability participants
Arm/Group | Surgery or Combination Chemotherapy, With/Without Radiotherapy
Number analyzed (Participants) | 183
Probability participants | 0.85 [0.78 to 0.89]

3. Secondary Outcome: Cure by Surgery Alone in Stage I Resected Patients
Description: To estimate the proportion of Stage I patients (with a single involved lymph node that is totally resected) who can be cured with surgery alone.
Time Frame: At 2 years
Population: Of 188 patients enrolled, five ineligible patients were excluded. 52 patients with Stage IA, single node LPHL were enrolled with a confirmed total resection (TR). The median follow up among the 39 censored patients is 56.3 months (range 3.9-107.4).
Measure: Number (95% Confidence Interval); unit: Probability participants
Arm/Group | Surgery or Combination Chemotherapy, With/Without Radiotherapy
Number analyzed (Participants) | 52
Probability participants | 0.82 [0.68 to 0.90]

4. Secondary Outcome: Cure by AV-PC x 3 or AV-PC x 3 + IFRT for Stage I Unresected, Stage I Resected Whose Disease Recurred, and Stage II Patients
Description: To estimate the proportions of Stage I unresected, Stage I resected (whose disease has recurred after observation), and Stage II LPHD patients who can be cured with AV-PC x 3, with IFRT for those who are not in a CR after chemotherapy.
Time Frame: At 5 years
Population: Of 188 patients enrolled, five ineligible patients were excluded. 136 patients received upfront AV-PC with or without RT per protocol. Of these 135 achieved CR with AV-PC and avoided RT. The median follow up among the 121 censored patients is 62.2 months (range 3.4-104.5).
Measure: Number (95% Confidence Interval); unit: Probability participants
Arm/Group | Surgery or Combination Chemotherapy, With/Without Radiotherapy
Number analyzed (Participants) | 135
Probability participants | 0.89 [0.82 to 0.93]

5. Secondary Outcome: Grade 3 or 4 Toxicity
Time Frame: Any time during chemoradiotherapy, up to the end of 3-cycles of AV-PC induction. Each cycle is 21 days.
Population: Eligible patients beginning AV-PC.
Measure: Number; unit: Participants
Arm/Group | Surgery or Combination Chemotherapy, With/Without Radiotherapy
Number analyzed (Participants) | 136
Participants | 26

ADVERSE EVENTS:
Description: For both Serious and Other: Adverse event incidence among 183 eligible participants. This is 188 enrolled less 5 that are ineligible. There were no (0) serious adverse events reported.
Arm/Group | Surgery or Combination Chemotherapy, With/Without Radiotherapy
Serious Adverse Events (participants affected / at risk) | 0/183
Other Adverse Events (participants affected / at risk) | 26/183
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery or Combination Chemotherapy, With/Without Radiotherapy (N=183)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
Catheter related infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.